CLINICAL TRIAL: NCT03071211
Title: Catheter Management After Pelvic Reconstructive Surgery: a Randomized Controlled Trial
Brief Title: Catheter Management After Pelvic Reconstructive Surgery
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Hartford Hospital (Other)
Responsible Party: Principal Investigator, Sarah Boyd, Fellow physician, Hartford Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: HHC-2016-0228
Record Dates: First submitted 2017-02-24; First posted 2017-03-06 (Actual); Last update posted 2019-02-04 (Actual); Status verified 2019-01

CONDITIONS: Urinary Retention Postoperative; Pelvic Organ Prolapse
Keywords: pelvic organ prolapse; urinary catheters
MeSH Terms: conditions — Pelvic Organ Prolapse

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (3):
- Plug-unplug Group (Experimental): Participants randomized to plug-unplug catheter management. Participants plug and unplug catheters when they feel urge to void or at least every 4 hours during the day. Participants are given the option to use a large drainage bag for convenience overnight.
  Interventions: Device: Plug-unplug catheter management
- Continuous Drainage Group (Active Comparator): Participants randomized to continuous drainage catheter management. Catheters are attached to a leg bag during the day and large drainage bag for convenience overnight.
  Interventions: Device: Continuous drainage catheter management
- Reference Group (No Intervention): Participants that do not fail inpatient voiding trial and go home without a catheter.

INTERVENTIONS:
Device: Plug-unplug catheter management — Transurethral catheter is plugged with a plastic cap and participants are taught to unplug during the day when they feel the urge to void or at least every 4 hours.
  Arms: Plug-unplug Group
Device: Continuous drainage catheter management — Transurethral catheter is attached to a continuous drainage bag.
  Arms: Continuous Drainage Group

SUMMARY:
This is a randomized controlled trial comparing plug-unplug catheter management, continuous drainage catheter systems and patients that do not get discharged with catheters after inpatient pelvic reconstructive surgery.

DETAILED DESCRIPTION:
This study will be a randomized controlled trial comparing plug-unplug (PUP) catheter management, continuous drainage (CD) catheter systems and patients that do not get discharged with catheters (reference) after pelvic reconstructive surgery. The primary objective of this study is to assess impact on activity. The secondary objectives are to compare the rate of urinary tract infection between the groups, duration of time (days) it takes for patients to resume normal voiding, impact on post-operative pain and satisfaction with surgery experience and post-operative recovery. The investigators hypothesize that patient activity/mobility one week after surgery between the two methods of managing the transurethral catheter will be different between arms. Subjects will be recruited at the Hartford Hospital Division of Female Pelvic Medicine and Reconstructive Surgery during preoperative consultation for pelvic reconstructive surgery with 1:1:1 assignment and randomization for PUP and CD groups only. Prior to surgery, baseline activity will be assessed using the Activity Assessment Scale, as well as postoperative expectations. Prior to hospital discharge, patients will undergo a postoperative voiding trial (PVT) per regular clinical practice. Upon failure of PVT, participants will be randomized 1:1 to one of two arms in which participants receive a catheter: PUP or CD. The investigator responsible for data collection will remain blinded to the treatment assignment throughout the study. Subjects who pass the PVT test and therefore do not require a catheter will be assigned to the reference arm (Arm C). Subjects will be followed after hospital discharge and assessed using the same pre- and post-operative questionnaires as participants randomized to the CD and PUP arms and will comprise the first 32 consenting patients who do not require a catheter.

Subjects randomized to CD will have a 16F transurethral catheter attached to a leg bag and receive teaching regarding home maintenance. Subjects randomized to PUP will have the same 16F transurethral catheter placed with a plastic plug and instructed to unplug and drain the catheter when they feel the urge to void, or at least every four hours throughout the day. Subjects in both groups will be provided a large bag for gravity-based drainage during the night. Subjects also will be encouraged to call the research team with any catheter-related questions or concerns including symptoms of urinary tract infection (UTI). Subjects with symptoms of UTI (e.g., dysuria, urgency, frequency, and/or hematuria) will be evaluated and treated per standard of care. All participants will then return for an office voiding trial (OVT) five to seven days after hospital discharge, following the same protocol as the PVT. At this time urinalysis will be obtained. Only those participants who endorse symptoms of UTI will have a urine specimen collected and sent for culture. This is in line with the current clinical practice by the investigators. Participants will be treated for UTI based on culture results or if there is high clinical suspicion at the time of office follow-up. Participants who fail the OVT will be discharged home with bladder drainage per standard of care and undergo routine follow-up until they pass a repeat voiding trial.

The subjects will complete a post-operative questionnaire assessing pain, impact on activity and satisfaction. Outcomes will be followed for up to six weeks after initial OVT if it is failed; however, no additional research-associated visits will be necessary from study participants beyond the initial office visit.

ELIGIBILITY:
Inclusion Criteria:

* Female
* Age 18-89
* Inpatient surgery
* surgery for pelvic organ prolapse with or without mid-urethral slings who fail initial voiding trial at the time of hospital discharge
* willing/able to provide written informed consent

Exclusion Criteria:

* male
* age < 18 or >89
* unwilling or unable to provide written informed consent
* undergoing outpatient surgery.
* planned postoperative catheter use
* discharged to a nursing facility or who are not candidates for the plug-unplug method for another reason (e.g., poor hand dexterity, paraplegia)
* suprapubic catheter placement
* procedures involving urethral bulking or Onabotulinum toxin A (Botox) injection
* procedures involving planned urethral or bladder surgery (e.g., fistula excision, mesh excision, excision of urethral diverticulum)
* procedures with only posterior vaginal repair
* presence of a neurologic condition affecting urinary function

Ages: 18 Years to 89 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Gender Based: Yes
Enrollment: 96 (Actual)
Dates: Start 2017-02-26 (Actual); Primary Completion 2018-12-07 (Actual); Study Completion 2019-01-31 (Actual)

PRIMARY OUTCOMES:
Activity Assessment Scale | Postoperative day 3-5
  Participants complete this 18-question survey preoperatively and 3-5 days postoperatively.

SECONDARY OUTCOMES:
Preoperative expectations | At the time of consent
  Patients complete a preoperative expectations survey prior to surgery.
Days until passing voiding trial | up to 6 weeks postoperatively
  Evaluate rates of passing voiding trial between arms
Urinary Tract infection | up to 6 weeks postoperatively
  Rates of urinary tract infection between arms

CONTACTS AND LOCATIONS:
Overall Officials: Sarah S Boyd, MD, Principal Investigator — Hartford Hospital; Elena Tunitsky-Bitton, MD, Principal Investigator — Hartford Hospital
Locations (1):
- Hartford Hospital, Hartford, Connecticut, United States

IPD SHARING:
Plan to Share IPD: Undecided
At this time, it is undecided if IPD will be made available to other researchers at the end of this study.

REFERENCES:
- [Derived] Boyd SS, O'Sullivan DM, Tunitsky-Bitton E. A Comparison of Two Methods of Catheter Management After Pelvic Reconstructive Surgery: A Randomized Controlled Trial. Obstet Gynecol. 2019 Nov;134(5):1037-1045. doi: 10.1097/AOG.0000000000003525. PMID 31599826